CLINICAL TRIAL: NCT05950165
Title: A Phase I/IIa, Open-label, Multicenter Study of the Safety and Efficacy of CHO-H01 As a Single Agent/Combined with Lenalidomide to Subjects with Refractory or Relapsed Non-Hodgkin's Lymphoma
Brief Title: A Study to Assess Safety and Efficacy of CHO-H01 As a Single Agent/Combined with Lenalidomide in Subjects with Refractory or Relapsed Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cho Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NHLHAT-001
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: CHO-H01; Anti-CD20 Antibodies; Large B-cell lymphoma; Follicular lymphoma; Glyco-engineered anti-CD20 antibody
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — Lenalidomide

STUDY DESIGN:
Intervention Model Description: 3+3 sequential cohort design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHO-H01 (Experimental): Dose escalation phase
  Phase 1:
  Five to six cohorts of escalating dose levels of CHO-H01 from 0.5mg/kg to 12 mg/kg.
  Interventions: Drug: CHO-H01
- CHO-H01+Lenalidomide (Experimental): Expansion phase with lenalidomide combination.
  Phase2a:
  Single cohort at Recommended Phase 2 Dose (RP2D) of CHO-H01.
  Interventions: Drug: CHO-H01 at RP2D; Drug: Lenalidomide

INTERVENTIONS:
Drug: CHO-H01 — Phase 1:
  Subjects will be administered intravenous (IV) infusion of assigned dose level of CHO-H01, once a week for 4 weeks (Cycle 1-28-Day cycle).
  From Cycle 2 onwards, on Day 1 of each subsequent 21-day cycle until disease progression (or a total of 6 cycles [19 weeks] of study).
  Arms: CHO-H01
Drug: CHO-H01 at RP2D — Subjects will be administered intravenous (IV) infusion of RP2D level of CHO-H01, once a week for 4 weeks (Cycle 1-28-Day cycle).
  From Cycle 2 onwards, on Day 1 of each subsequent 28-day cycle until disease progression (or a total of 6 cycles [19 weeks] of study).
  Arms: CHO-H01+Lenalidomide
Drug: Lenalidomide — Subjects will receive oral lenalidomide 20 mg once daily from Day 1 to Day 21 per 28-day cycle.
  Arms: CHO-H01+Lenalidomide

SUMMARY:
This is a 2-part study. Part 1/Phase 1 of the study will be conducted to determine the safety and tolerability of CHO-H01 in subjects with relapsed/refractory CD20+ non-Hodgkin's lymphoma. It will also determine maximum tolerated dose (MTD) and recommended phase II dose (RP2D).

Part 2/Phase 2a will assess the anticancer activity and safety of CHO-H01 plus lenalidomide in subjects with low-grade relapsed/refractory CD20+ non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Phase I FIH study includes subjects with relapsed/refractory CD20 + non-Hodgkin's lymphoma, who may benefit from treatment with CHO-H01. In Phase I of the study, the first 2 cohorts will follow a 2-step modified accelerated titration dose escalation design and subsequent cohorts will follow a standard 3+3 dose escalation design.

The investigational medicinal product, CHO-H01, will be administered via IV infusion once weekly for 4 weeks in Cycle 1 and then once only (on Day 1) in each subsequent 21-day cycle until disease progression or for up to 6 cycles (19 weeks) of treatment.

Once the MTD/RP2D has been confirmed, Phase IIa of the study will be initiated. The purpose of Phase IIa is to assess anticancer activity and safety of CHO-H01 plus lenalidomide in low-grade relapsed/refractory CD20 + non Hodgkin's lymphoma, including follicular lymphoma (Grades 1-3a), marginal zone lymphoma, and small lymphocytic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of >12 weeks.
* Body mass index of 18 to 32 kg/m2.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Phase I: Have histologically (laboratory test) confirmed CD20 + non-Hodgkin's lymphoma according to the World Health Organization's 2016 classification:

  1. Low grade lymphoma: follicular lymphoma (Grades 1-3a), marginal zone lymphoma, small lymphocytic lymphoma;
  2. Other lymphoma: DLBCL (NOS: to include germinal center B-cell-like [GCB] and activated B-cell-like [ABC]), follicular lymphoma Grade 3b, mantle cell lymphoma; primary mediastinal large B-cell lymphoma.
* Phase IIa: Histologically confirmed CD20 + non-Hodgkin's lymphoma according to the World Health Organization's 2016 classification, only low grade lymphoma: follicular lymphoma (Grades 1-3a), marginal zone lymphoma, small lymphocytic lymphoma.
* Have at least one measurable lesion that is at least 1.5 cm in its largest dimension.
* Off treatment for 30 days from last anti-CD20 infusion until planned administration of CHO-H01.
* If no original sample is available, is willing and able to provide an adequate tumor biopsy sample at Screening.
* Have adequate cardiac function: without clinically significant and/or uncontrolled heart disease.
* Must be sterile, or have a monogamous partner who is surgically sterile, or at least 2 years postmenopausal, or be committed to use an acceptable form of birth control for the duration of the study (male), and for the duration of the study and for 3 months following the last CHO-H01 administration (female).

Exclusion Criteria:

* Must not have a history of egg allergy or allergic reactions to any component of CHO-H01.
* Must not have any known or current illnesses (such as autoimmune disease, unless well controlled or resolved), infection, or other condition that could limit study compliance or interfere with assessments.
* Subjects who have received anti-programmed death-ligand 1 (PD-L1), programmed cell death 1 (PD-1), or cytotoxic T-lymphocyte associated protein 4 (CTLA-4) therapy.
* Subjects who have completed an autologous stem cell transplant within 100 days prior to CHO-H01 therapy or an allogeneic stem cell transplant.
* Subjects with known hepatitis B surface antigen (HBsAg) seropositive or known or suspected active hepatitis C infection with detectable viral load.
* Subjects with known human immunodeficiency virus (HIV) infection
* Subjects who have had radiation therapy, major surgical procedure or live vaccinations within 28 days prior to CHO-H01 administration.
* Subjects with a history of type I hypersensitivity or anaphylactic reactions to murine proteins or to previous infusions of CD20 monoclonal antibodies.
* Subjects who have received (or are receiving) systemic corticosteroids:

  1. At a daily dose higher than 15 mg prednisone or equivalent within 14 days prior to the first administration of CHO-H01;
  2. Topical, inhaled, nasal, and ophthalmic steroids are allowed.
* Inadequate bone marrow, hepatic or renal function.
* Subjects with a history of seizure disorder.
* Subjects who are pregnant or breast feeding.
* Subjects with any contraindications to lenalidomide (Only for phase IIa).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AE) | Through study completion, approximately 16 months
  To assess the safety and tolerability of CHO-H01 as a single agent in subjects with relapsed/refractory CD20 + non-Hodgkin's lymphoma and CHO-H01 plus lenalidomide in subjects with low-grade relapsed/refractory CD20 + non-Hodgkin's lymphoma.
Number of subjects with dose-limiting toxicities | Through study completion, approximately 16 months
  All AEs and toxicities are evaluated based on the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 5.0. The 5 general grades are Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-threatening or disabling, and Grade 5: Death (outcome of AE).
Objective Response Rate | Through study completion, approximately 16 months
  Objective response rate (ORR) is the proportion of subjects with a best overall response of complete response (CR) or partial response (PR). ORR will be measured based on Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.
Best overall response | Through study completion, approximately 16 months
  The best overall response (CR, PR, stable disease [SD], or progressive disease [PD]) is defined as the best response across all time points.

SECONDARY OUTCOMES:
Serum concentration of CHO-HO1 | Through study completion, approximately 16 months
  To characterize the PK of CHO-H01.
Serum Antidrug antibody (ADA) concentration | Through study completion, approximately 16 months
  To investigate the immunogenicity of CHO-H01 alone and in combination with lenalidomide, using a validated bridging ADA assay.
Clinical benefit rate | Through study completion, approximately 16 months
  The clinical benefit rate (CBR) is the proportion of subjects who achieve CR, PR, and durable SD (SD ≥12 weeks) based on the Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.
Time to event endpoints of time to progression (TTP) | Through study completion, approximately 16 months
  Time to progression is the time from the date of first study dose to disease progression, evaluated using Modified (not using PET imaging)Lugano Revised Criteria for Response assessment.
Duration of stable disease | Through study completion, approximately 16 months
  Duration of SD defined as the time interval, in the absence of either CR or PR, will be calculated between the date of the first CHO-H01 administration and the date of disease progression or death for any cause, whichever occurs earlier; based on the Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.
Progression-free survival | Through study completion, approximately 16 months
  Progression-free survival (PFS) is the time from the date of first study dose to disease progression or death whichever occurs first in subjects, evaluated using Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.
Duration of response | Through study completion, approximately 16 months
  Duration of response for responders (CR or PR) is the time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier; based on the Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.
Overall survival | Through study completion, approximately 16 months
  The overall survival (OS) is the time from the date of the first study dose to the date of death (any cause), evaluated using Modified (not using PET imaging) Lugano Revised Criteria for Response assessment.

CONTACTS AND LOCATIONS:
Locations (8):
- Renovatio Clinical, The Woodlands, Texas, United States
- Taiwan (7):
  - Tri-Service General Hospital - Neihu Branch - Hematology, Taipei, Taipei
  - Taipei Medical University - Shuang Ho Hospital - Oncology, New Taipei City, Taipei Special Municipality
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Hematology and Oncology - Hematology and Oncology, Taoyuan District, Taoyuan
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital - Hemato-Oncology, Kaohsiung City
  - China Medical University Hospital - Hematology/Oncology - Taichung, Taichung
  - National Cheng Kung University Hospital - Internal Medicine, Tainan
  - National Taiwan University Hospital - Hematology And Oncology, Taipei

IPD SHARING:
Plan to Share IPD: No